CLINICAL TRIAL: NCT03976349
Title: A Phase 1 Single- and Multiple-Ascending-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of BIIB094 Administered Intrathecally to Adults With Parkinson's Disease
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BIIB094 in Adults With Parkinson's Disease
Acronym: REASON
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 254PD101; 2018-002995-42 (EudraCT Number)
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — BIIB094

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part A (SAD): BIIB094 Dose 1 (Experimental): Participants will receive a single IT injection of BIIB094 during Part A [Single Ascending Dose (SAD)].
  Interventions: Drug: BIIB094
- Part A (SAD): BIIB094 Dose 2 (Experimental): Participants will receive a single IT injection of BIIB094 during Part A (SAD).
  Interventions: Drug: BIIB094
- Part A (SAD): BIIB094 Dose 3 (Experimental): Participants will receive a single IT injection of BIIB094 during Part A (SAD).
  Interventions: Drug: BIIB094
- Part A (SAD): BIIB094 Dose 4 (Experimental): Participants will receive a single IT injection of BIIB094 during Part A (SAD).
  Interventions: Drug: BIIB094
- Part A (SAD): BIIB094 Dose 5 (Experimental): Participants will receive a single IT injection of BIIB094 during Part A (SAD).
  Interventions: Drug: BIIB094
- Part A (SAD): BIIB094 Dose 6 (Experimental): Participants will receive a single IT injection of BIIB094 during Part A (SAD).
  Interventions: Drug: BIIB094
- Part B (MAD): BIIB094 Dose 1 (Experimental): Participants will receive a single IT injection of BIIB094 on multiple days during Part B [Multiple Ascending Dose (MAD)].
  Interventions: Drug: BIIB094
- Part B (MAD): BIIB094 (Non LRRK2) Dose 2 (Experimental): Participants [Non leucine-rich repeat kinase 2 (Non LRRK2)] will receive a single IT injection of BIIB094 on multiple days during Part B (MAD).
  Interventions: Drug: BIIB094
- Part B (MAD): BIIB094 (LRRK2) Dose 2 (Experimental): Participants (LRRK2) will receive a single IT injection of BIIB094 on multiple days during Part B (MAD).
  Interventions: Drug: BIIB094
- Part B (MAD): BIIB094 (Non LRRK2) Dose 3 (Experimental): Participants (Non LRRK2) will receive a single IT injection of BIIB094 on multiple days during Part B (MAD).
  Interventions: Drug: BIIB094
- Part B (MAD): BIIB094 (LRRK2) Dose 3 (Experimental): Participants (LRRK2) will receive a single IT injection of BIIB094 on multiple days during Part B (MAD).
  Interventions: Drug: BIIB094
- Part A (SAD): Matching Placebo (Placebo Comparator): Participants will receive matching placebo during Part A [Single Ascending Dose (SAD)].
  Interventions: Drug: Placebo
- Part B (MAD): Matching Placebo (Placebo Comparator): Participants will receive matching placebo on multiple days during Part B (MAD).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB094 — Administered as specified in the treatment arm.
  Arms: Part A (SAD): BIIB094 Dose 1; Part A (SAD): BIIB094 Dose 2; Part A (SAD): BIIB094 Dose 3; Part A (SAD): BIIB094 Dose 4; Part A (SAD): BIIB094 Dose 5; Part A (SAD): BIIB094 Dose 6; Part B (MAD): BIIB094 (LRRK2) Dose 2; Part B (MAD): BIIB094 (LRRK2) Dose 3; Part B (MAD): BIIB094 (Non LRRK2) Dose 2; Part B (MAD): BIIB094 (Non LRRK2) Dose 3; Part B (MAD): BIIB094 Dose 1
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Part A (SAD): Matching Placebo; Part B (MAD): Matching Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of single and multiple doses of BIIB094 administered via intrathecal (IT) injection to participants with Parkinson's Disease (PD). The secondary objective of this study is to evaluate the pharmacokinetic (PK) profile of BIIB094.The study is open for PD patients with verified presence or absence of variations in the leucine-rich repeated kinase 2 (LRRK2) gene, but also for patients without any verified PD-related genetic variant.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local participant privacy regulations.
* Diagnosed with PD within 7 years at the time of initial enrollment (i.e., at time of SAD enrollment for rollover participants), without major motor fluctuations or dyskinesia that may interfere with study treatment and assessments in the opinion of the investigator after consultation with the Sponsor.
* Modified Hoehn and Yahr Stage ≤ 3.

Key Exclusion Criteria:

* Montreal Cognitive Assessment (MoCA) score less than (<) 23, dementia, or other significant cognitive impairment that, in the opinion of the Investigator, would interfere with study evaluation.
* History of any brain surgery for PD or a history of focused ultrasound treatment at any time; or history of neuromodulation procedures.
* Transient ischemic attack or stroke or any unexplained loss of consciousness within 1 year before Screening.
* History of unstable angina, myocardial infarction, chronic heart failure, or clinically significant conduction abnormalities within 1 year before Screening.
* Poorly controlled diabetes mellitus, as defined by having dosage adjustment of diabetic medication within 3 months before dosing (Day 1) or glycosylated hemoglobin value greater than or equal to (≥) 8 percent (%) at Screening.
* History or positive test result at Screening for human immunodeficiency virus.
* History or positive test result at Screening for hepatitis C virus antibody.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Part A: Screening (Day -42) up to Day 85, Part B: Screening (Day -77) up to Day 253
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); however, this does not include an event that, had it occurred in a more severe form, might have caused death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; is a medically important event.

SECONDARY OUTCOMES:
Serum Concentrations of BIIB094 | Part A: pre-dose through Day 57, Part B: pre-dose through Day 169
Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUCinf) of BIIB094 | Part A: pre-dose through Day 57, Part B: pre-dose through Day 169
Area Under the Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast) of BIIB094 | Part A: pre-dose through Day 57, Part B: pre-dose through Day 169
Maximum Concentration (Cmax) of BIIB094 | Part A: pre-dose through Day 57, Part B: pre-dose through Day 169
Time to Reach Maximum Concentration (Tmax) of BIIB094 | Part A: pre-dose through Day 57, Part B: pre-dose through Day 169
Terminal Elimination Half-Life (t1/2) of BIIB094 | Part A: pre-dose through Day 57, Part B: pre-dose through Day 169

CONTACTS AND LOCATIONS:
Locations (18):
- United States (7):
  - Northwestern University PD and Movement Disorders Center, Chicago, Illinois
  - Quest Research Institute, Farmington Hills, Michigan
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Alliance for Multispecialty Research, Knoxville, Tennessee
  - Inland Northwest Research, Spokane, Washington
- Canada (2):
  - Research Site, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Sourasky Medical Center, Tel Aviv, Israel
- Norway (2):
  - Neuro-SysMed Center, Bergen
  - St. Olav University Hospital, Trondheim
- Spain (5):
  - Laboratorios de Investigación Biocruces 3., Hospital de Cruces, Barakaldo, Bizkaia
  - Hospital General de Catalunya, Barcelona, Vizcaya
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Research Site, Seville
- Queen Square (Neurology) CRF Site Institute of Neurology & the National Hospital for Neurology and Neurosurgery UCLH, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No